CLINICAL TRIAL: NCT05333185
Title: The Effect of Mobile Application Robot Developed for Pediatric Diabetes Management on Children With Diabetes Mellitus (DM)
Brief Title: The Effect of Mobile Application on the Pediatric Diabetes Management
Acronym: DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Murat Bektaş, Prof. Dr., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: NECMETTİN ERBAKAN U
Record Dates: First submitted 2022-03-21; First posted 2022-04-18 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 1; Child; Adolescent
Keywords: Type 1 Diabetes,; Children,; Self-Management,; Mobile Application
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: The child with type 1 diabetes will be divided into two as the experimental and control group. Children in the experimental group will be informed about the diabot application and how they will use the application to manage their disease processes. Children/adolescents in the study group and their parents will be evaluated 5 times, once every 3 months, through data collection tools. Data will be collected from the children/adolescents in the control group and their parents by means of pre-test and data collection tools 5 times, once every 3 months. If the training is found effective after the study is completed, similar training will be given to the control group via the mobile application.
Who Masked: Participant, Investigator
Masking Description: single bilinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Children in the experimental group will be informed about the diabot application and how they will use the application to manage their disease processes. Children/adolescents in the study group and their parents will be evaluated 5 times, once every 3 months, through data collection tools. Data will be collected from the children/adolescents in the control group and their parents by means of pre-test and data collection tools 5 times, once every 3 months.
  Interventions: Behavioral: DİABOT (mobile application robot )
- Control group (No Intervention): The control group will recieve standard diabetes treatment without any training intervention

INTERVENTIONS:
Behavioral: DİABOT (mobile application robot ) — DİABOT (mobile application robot ) Thanks to the trainings given through the mobile application robot developed for pediatric diabetes management, it is aimed to have an effect on the quality of life, diabetes self-management and physiological parameter levels of children with Type
  1 diabetes, and to easily obtain the information they need even when they cannot come to the outpatient clinic. In addition, thanks to the application robot, he will be able to create his own exercise program and determine his diet.
  Arms: Experimental group

SUMMARY:
Type 1 DM; It is a chronic metabolic disease that develops as a result of the destruction of pancreatic ß cells, which are responsible for insulin production.

Although type 1 DM can occur at any age, the highest incidence is seen between the ages of 10-14. Especially in this age group (7-15 years), who are more social than the previous period with the emergence of diabetes symptoms, both physical restrictions and limitations in their emotional and social functionality permanently change the lives of children with diabetes. According to the International Diabetes Federation (IDF) 2019 data, it is estimated that the patients with Type 1 diabetes in the world are 1,110,100 children/adolescents. This number is increasing each year, and it is estimated that approximately 98,200 children and adolescents under the age of 15 are diagnosed with Type

1 diabetes each year. It is seen that there is an increase in the number of cases in young children in high-risk groups. Therefore, early diagnosis and initiation of treatment is a necessary step. The basic elements of type 1 diabetes treatment are; diabetes education, nutrition, exercise, insulin, blood sugar monitoring and psychosocial counseling. Recently; It is seen that the use of technology in children with diabetes has increased thanks to the opportunity to access information at any time, to choose the information according to one's own needs, to receive service when it is ready, to reduce costs in health, and to be educated at home due to limitations. Taking measures to prevent worsening of glycemic regulation and weight gain in patients with diabetes, especially in situations that cause social isolation such as pandemics, monitoring and management of patients with diabetes during the social isolation process, and enabling patients to access the information they need in a short time are of great importance in terms of diabetes tables. When the literature is examined, it is seen that there are many pages and mobile applications related to this. In this study, it is aimed to improve the self-management of children/adolescents with a mobile application that can be accessed from any device suitable for today. For this, it is aimed to create a mobile application that includes all sub-dimensions of diabetes self-management and contains content that other applications do not have.

DETAILED DESCRIPTION:
Type 1 DM; It is a chronic metabolic disease that develops as a result of the destruction of pancreatic ß cells, which are responsible for insulin production.

Although type 1 DM can occur at any age, the highest incidence is seen between the ages of 10-14. Especially in this age group (7-15 years), who are more social than the previous period with the emergence of diabetes symptoms, both physical restrictions and limitations in their emotional and social functionality permanently change the lives of children with diabetes. According to the International Diabetes Federation (IDF) 2019 data, it is estimated that the patients with Type 1 diabetes in the world are 1,110,100 children/adolescents. This number is increasing each year, and it is estimated that approximately 98,200 children and adolescents under the age of 15 are diagnosed with Type

1 diabetes each year. It is seen that there is an increase in the number of cases in young children in high-risk groups. Therefore, early diagnosis and initiation of treatment is a necessary step. The basic elements of type 1 diabetes treatment are; diabetes education, nutrition, exercise, insulin, blood sugar monitoring and psychosocial counseling. Recently; It is seen that the use of technology in children with diabetes has increased thanks to the opportunity to access information at any time, to choose the information according to one's own needs, to receive service when it is ready, to reduce costs in health, and to be educated at home due to limitations. Taking measures to prevent worsening of glycemic regulation and weight gain in patients with diabetes, especially in situations that cause social isolation such as pandemics, monitoring and management of patients with diabetes during the social isolation process, and enabling patients to access the information they need in a short time are of great importance in terms of diabetes tables. When the literature is examined, itis seen that there are many pages and mobile applications related to this. In this study, it is aimed to improve the self-management of children/adolescents with a mobile application that can be accessed from any device suitable for today. For this, it is aimed to create a mobile application that includes all sub-dimensions of diabetes self-management and contains content that other applications do not have. When the previously developed mobile application programs and their features were investigated for this study, a search was made with the keywords "Diabetes", "Type 1 DM", "T1DM" in the Play Store and App Store, and a total of 70 applications were reached. When participants look at the features of these applications, it is seen that the educational contents are specially designed for adults and most of them are in foreign languages. Blood sugar monitoring, exercise duration and type, carbohydrate levels and blood pressure values can be followed through programs, only 9 of which are in Turkish. When these applications are compared with the mobile application robot that participants plan to develop for diabetes management; Being the first Turkish mobile application robot specially designed for children with diabetes, having age-specific content, having a whatsapp business api application within the program, where they can reach the healthcare professional 24/7, sending personalized daily tips, synchronized use of the child and parent, having a voice response system, game-based It is among the privileges of the program that it includes training, digital technologies in health", "Science, Technology and Society", "Information and information technologies", being among the priority areas, and meeting the 11th Development targets of the Grand National Assembly of Turkey. In addition to contributing to the economy of our country by preventing acute and chronic complications in children, increasing the quality of life of children, bringing a new application to the field of health technologies, contributing to the fields of child health and diseases and pediatric health and diseases nursing, this robot participants will make for pediatric patients with diabetes. It is foreseen that the publications and presentations in the scientific fields will increase the scientific visibility and prestige of our country and will have a widespread impact at the international level.

ELIGIBILITY:
Inclusion Criteria:

* Be in the 7-12 age range
* Understanding and speaking Turkish
* No vision or hearing problems
* Having been diagnosed with Type 1 Diabetes Mellitus at least six months ago
* Parents and children must have an internet connection, computer, smartphone or tablet to use the Diabot application

Exclusion Criteria:

* The children who will participate in the research have another chronic disease together with diabetes,

  * The children who will participate in the study have a neurological disease together with diabetes,
  * No internet connection and no smartphone or tablet,
  * Not having the ability to use the application.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Diabetes Self-Management Scale for Children and parents mean score | 3- 15 months
  The mean scores of the diabetes self-management scale for children and parents of the intervention and control groups were to be compared at the 3rd, 6th, 9th and 12th months.
Quality of life Scale for Children With Diabetes Mellitus Mean Score | 3- 15 months
  The mean scores of the diabetes Quality of Life scale for children of the intervention and control groups were to be compared at the 3rd, 6th, 9th and 12th months.
HbA1c Levels | 3- 15 months
  HBA1c levels of intervention and control groups will be compared at 3rd, 6th, 9th and 12th months.
Blood Glucose Levels | 3- 15 months
  Blood Glucose Levels of intervention and control groups will be compared at 3rd, 6th, 9th and 12th months.

SECONDARY OUTCOMES:
the increase in the number of children exercising regularly compared to the baseline, according to the physical exercise registration form. | 3-15 months
  Regular exercise status of the intervention and control groups at the 3rd, 6th, 9th and 12th months will be compared.
Number of hospitalizations and emergency department admissions | 3-15 months
  The number of hospitalizations and admissions to the emergency department in the 3rd, 6th, 9th and 12th months of the intervention and control groups will be compared. Applications will be determined by hospitalization and emergency service application form.
  hyperglycemia (high blood sugar)
Regulating the Nutrition of Children according to their blood sugar level | 3-15 months
  regulating the nutrition of children according to their blood sugar level using the mobile application

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University Medical Faculty Hospital, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The researcher at Necmettin Erbakan University will assist in data collection.